CLINICAL TRIAL: NCT03699592
Title: Reach Home and Read
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment.
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: Pro00086166
Record Dates: First submitted 2018-01-24; First posted 2018-10-09 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Literacy
MeSH Terms: conditions — Literacy

STUDY DESIGN:
Intervention Model Description: time series prospective cohort and comparison group design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention)
- Reach Home and Read (Experimental): This arm will receive the Reach Home and Read early literacy intervention
  Interventions: Behavioral: Reach Home and Read Toolkit

INTERVENTIONS:
Behavioral: Reach Home and Read Toolkit — The toolkit currently includes one age-appropriate book along with a set of educational pamphlets explaining the importance home literacy. These educational materials focus on appropriate literacy milestones and descriptions of how parents can engage with their children around books. In addition, we will create an information sheet outlining zipcode-specific community literacy resources, including location and information on how to access the library, where to obtain low-cost books, and a schedule of literacy promotion activities in their community (e.g. community reading sessions). All materials will also be translated into Spanish by a certified interpreter, and will be reviewed to ensure that they are written at a fifth grade reading level. Additionally, EDCI families receiving this intervention will also receive an additional new book at each home visit conducted during the study period.
  Arms: Reach Home and Read

SUMMARY:
This will be a time series prospective cohort and comparison group design to evaluate the effect on home literacy environments of the Reach Home and Read intervention as compared to standard programming provided by home visiting staff. The intervention will consist of staff training for East Durham Children's Initiative (EDCI) early childhood staff and the provision of an age appropriate book at their home visits.

The control group will be children receiving the current EDCI home visiting programming. The intervention group will receive standard EDCI programming and the Reach Home and Read intervention administered by the EDCI early childhood home visiting staff.

The standardized StimQ home literacy assessment tool will be used to measure changes in the home literacy environment. Additionally, a qualitative portion of this study will inform future research and tool-kit design. The design is a qualitative descriptive study that utilizes the methodologies of focus groups for data collection.

DETAILED DESCRIPTION:
The ROR-h Toolkit: The toolkit currently includes one age-appropriate book along with a set of educational pamphlets explaining the importance home literacy. These educational materials focus on appropriate literacy milestones and descriptions of how parents can engage with their children around books. The investigators will conduct pre-study, preliminary testing of the toolkit among at least five families and EDCI staff participating in EDCI's Parent Café, and incorporate changes. In addition, the investigators will create an information sheet outlining zipcode-specific community literacy resources, including location and information on how to access the library, where to obtain low-cost books, and a schedule of literacy promotion activities in their community (e.g. community reading sessions). All materials will also be translated into Spanish by a certified interpreter, and will be reviewed to ensure that they are written at a fifth grade reading level using web-based technology (Microsoft Word). Additionally, EDCI families receiving this intervention will also receive an additional new book at each home visit conducted during the study period.

The baseline cohort of 50 families will be recruited from families receiving EDCI early childhood home visits. Families will be approached by EDCI staff and will be asked whether they are interested in being contacted about participation in the study. Because our intervention includes children aged 6-12 months, EDCI staff will approach all families with children aged 5-11 months who participate in the early childhood program. If a family agrees to be contacted, a trained research assistant will contact and consent the family by phone. Once consent is obtained, baseline demographic information will be collected via REDCap. This information will include patient age, patient race, number of children in the family, parent age, parent education, insurance, and primary language spoken in the home. Baseline StimQ assessment data will also be collected and entered into REDCap. When possible, information will be entered into REDCap electronically by the family from their own electronic device. When this is not possible, the research assistant will collect this data electronically in person or by phone.

Once the family is enrolled and baseline StimQ data has been collected, EDCI staff will continue to provide their standard home visiting services. After three months, families will be sent a follow up StimQ assessment to be completed electronically via REDCap. If the family does not complete this follow up, they will be contacted by the research assistant to complete this follow up at two week intervals for 6 weeks.

Once the baseline cohort has completed their 3 month study period, EDCI staff will receive tool-kit training. The study PI (Erickson) will conduct a one-hour training session with all EDCI home visitors. The training will cover the importance of literacy in health and wellness, the impact of exposure to books and reading in children and how this affects their social and emotional development, and how to implement this model of teaching in their home visit. EDCI home visitors will also complete online modules validated by ROR.

Once training is complete, recruitment and enrollment for the intervention group will begin. Families will be approached by EDCI staff and will undergo the same recruitment and enrollment procedure as above. We plan to enroll and additional 50 families in this cohort. Demographic information and baseline StimQ data will be conducted as above. Once families are enrolled, EDCI staff will provide the literacy toolkit described above at the next scheduled home visit and engage actively with the family around the importance of early literacy using the kit as a tool to model positive interactions. EDCI staff will provide an additional book at each scheduled monthly visit over the next 3 months and an additional fact sheet outlining age appropriate literacy milestones at 3 months. At the completion of the 3 month intervention period, families will be sent a follow up StimQ assessment to be completed electronically via REDCap. If the family does not complete this follow up, they will be contacted by the research assistant to complete this follow up at two week intervals for 6 weeks. Families will also be provided with acceptability surveys at this time.

For the qualitative portion of this study, 15-20 key informants will be recruited. Interviews and/or focus groups will be held at the EDCI office and facilitated by a member of the DOCR research services team versed in qualitative data collection and analysis. The facilitator will utilize a guide during group discussions and/or interviews which will serve to structure conversations around relevant questions. Study participants will be asked to answer a few demographic questions before sharing experiences and perspectives. The groups and/or interviews will be recorded on a secure digital recorder; the audio file will be uploaded immediately to a secure Duke server. Individual participation will last approximately 1 hour and refreshments will be provided.

ELIGIBILITY:
Inclusion Criteria:

* Families who live within the EDCI zone Families who can read and write in English and/or Spanish Families with children aged 6 months to 12 months at the time of enrollment Children born at >37 weeks gestation

Exclusion Criteria:

* Parent with severe medical or mental health condition limiting ability to attend appointments Child with severe medical or mental health condition limiting ability to attend appointments or participate in behavioral therapies Parent and child plan to move out of state in the next 6 months, or plan to live in another state for 2 months or longer within the next 6 months (ex., summer vacation).

Ages: 6 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2019-04-02 (Actual); Study Completion 2019-04-02 (Actual)

PRIMARY OUTCOMES:
Home Literacy Environment | 6 months
  Stim-Q scores
Number of participants that enjoyed the program measured by a survey | Up to 6 months
Number of participants that liked the books provided in the program measured by a survey | Up to 6 months
Number of participants that stated they liked the information provided about early literacy measured by a survey | Up to 6 months
Number of staff members that stated they liked the program as measured by a survey | Up to 6 months
Number of staff members that stated the program was easy to administer as measured by a survey | Up to 6 months
Number of staff members that stated they liked the books provided in the program measured by a survey | Up to 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Duke Children's Primary Care, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided